CLINICAL TRIAL: NCT00298155
Title: Maximal Suppression of the Androgen Axis in Clinically Localized Prostate Cancer
Acronym: TAPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: GlaxoSmithKline (Industry); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Bruce Montgomery, Professor, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28741; FHCRC-05026 (Other: Cancer Consortium IRB); 05-8538-V 01 (Other: U. of Washington IRB (old application number)); 28741-A (Other: U. of Washington IRB (application number); dual review); 01253 (Other: VA Puget Sound Health Care System IRB (current))
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Cancer; Prostate Neoplasms
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms | interventions — Goserelin; Dutasteride; bicalutamide; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Active Comparator): Goserelin + dutasteride
  Interventions: Drug: goserelin with dutasteride
- Group 2 (Active Comparator): Bicalutamide for one week, begin goserelin plus dutasteride, continue bicalutamide for the full 12 weeks
  Interventions: Drug: goserelin with bicalutamide and dutasteride
- Group 3 (Active Comparator): Begin bicalutamide for one week, goserelin injection; begin dutasteride, ketoconazole (and replacement hydrocortisone), continue bicalutamide for the full 12 weeks
  Interventions: Drug: goserelin with bicalutamide and dutasteride and ketoconazole

INTERVENTIONS:
Drug: goserelin with dutasteride — Bicalutamide 50 mg qd for one week, inject goserelin 10.8 mg (3-month depot) and begin dutasteride 3.5 mg qd; continue bicalutamide for one more week.
  Arms: Group 1
Drug: goserelin with bicalutamide and dutasteride — Bicalutamide 50 mg qd for one week, inject goserelin 10.8 mg (3-month depot) and begin dutasteride 3.5 mg qd.
  Arms: Group 2
Drug: goserelin with bicalutamide and dutasteride and ketoconazole — Bicalutamide 50 mg qd for one week, inject goserelin 10.8 mg (3-month depot), begin dutasteride 3.5 mg qd and ketoconazole 200 mg tid (with hydrocortisone 30 mg).
  Arms: Group 3

SUMMARY:
Prostate cancer (CaP) is the most commonly diagnosed cancer among males in the U.S. and the second leading cause of cancer-related mortality. More than 230,000 men will be diagnosed with prostate cancer in the USA this year and more than 30,000 will die of this disease.

Androgen deprivation, the elimination of testosterone and its active metabolites, remains the single most effective intervention available for the treatment of advanced prostate carcinoma. This is usually achieved by surgical removal of the testes (orchiectomy), by suppressing production of testosterone (LHRH agonists) and/or by blocking the androgens at receptor sites (antiandrogens). Unfortunately, androgen suppression does not cure the disease. Most patients progress within 0-5 years, and all patients ultimately progress if the cancer is not eliminated during initial therapy (usually prostatectomy or radiation).

Hormone suppression treatment eliminates the detectable levels of testosterone in the blood. However, the testosterone levels in tissue remain high enough to stimulate androgen receptors. Overexpression of androgen receptors is present in all cell lines which demonstrate "androgen independence," i.e., are resistant to androgen-suppressive therapy.

Approximately 95% of testosterone is supplied by the testes, with the remaining 5% supplied by the adrenal glands. The presumption that standard androgen deprivation achieves the optimal level of androgen suppression for patients is based on the levels of androgen which result from orchiectomy. However, because adrenal androgen levels are unaffected by standard modes of androgen deprivation, 5% of the body's testosterone remains despite hormone therapy.

The hypothesis of this study is that more effective suppression of the androgen axis through elimination of adrenal androgens and more effective suppression of testosterone metabolites will lower intraprostatic androgen levels, minimizing activation of the androgen receptor and augmenting natural cell death (apoptosis). The investigators propose to test this hypothesis by administering neoadjuvant (pre-surgery) androgen deprivation therapy of different types before prostatectomy for patients with clinically localized prostate cancer. The investigators will assay serum and intraprostatic androgen levels, while assessing relative levels of apoptosis of normal and malignant tissue.

DETAILED DESCRIPTION:
Androgen deprivation has been the principal means of controlling advanced prostate cancer, but does not cure the disease and all patients ultimately progress if the tumor is not eliminated with definitive local therapy. It has been demonstrated that despite androgen deprivation with LHRH agonists or orchiectomy, prostate tissue and prostate cancer maintain levels of androgens which are more than adequate to stimulate the androgen receptor. These levels of androgen may continue to stimulate the receptor and allow both survival of tumor cells and induction of resistance by overexpression of the receptor. The presumption that standard androgen deprivation achieves the optimal level of androgen suppression for patients is based on the levels of androgen achieved with castration, which achieves relatively short term control of cancer in the majority of patients. The hypothesis of this study is that more effective suppression of the androgen axis through elimination of adrenal androgens and more effective suppression of conversion to dihydrotestosterone will lower intraprostatic androgen levels, minimizing activation of the androgen receptor and augmenting apoptosis. We propose to test this hypothesis in a prospective, randomized trial, administering neoadjuvant androgen deprivation therapy of different types prior to radical prostatectomy for patients with clinically localized prostate cancer for 3 months.

Plan of therapy

Patients with clinically localized (cT1-T2) prostate cancer, at intermediate-high risk for relapse who are candidates for radical prostatectomy will be treated with one of three regimens:

* Goserelin with dutasteride
* Goserelin with bicalutamide and dutasteride
* Goserelin with bicalutamide and dutasteride and ketoconazole

Patients will undergo radical prostatectomy 3 months after initiation of treatment.

Preoperative and intraoperative biopsies of the prostate gland will be utilized for analysis of prostatic hormones, gene expression and apoptosis.

ELIGIBILITY:
Inclusion Criteria:

1. Men 18 years or older with a histologic diagnosis of clinically localized prostate cancer prior to radical prostatectomy as defined by:

   * Clinical stage T1-T2b
   * Prostate specific Antigen (PSA) less than 20
   * Gleason score 7-10
2. Patient's tumor must be considered surgically resectable .
3. Eastern Cooperative Group (ECOG) performance status of 0-1.
4. Life expectancy greater than 2 years.
5. Able to understand and give informed consent.
6. Laboratory values must be within specified limits.

Exclusion Criteria:

1. Patients with locally advanced or high risk disease not meeting the criteria defined above.
2. Patients who have a total testosterone less than 280 ng/dL.
3. Patients who are receiving any other investigational therapy.
4. Patients with an active serious infection or other serious underlying medical condition.
5. Dementia or significantly altered mental status that would prohibit the understanding and/or giving of informed consent.
6. Histologic evidence of small cell carcinoma of the prostate.
7. Patients who are currently receiving active therapy for other neoplastic disorders.
8. Patients who are receiving any androgens, estrogens or progestational agents.
9. Patients who are taking drugs or herbal supplements which affect androgen metabolism (e.g., spironolactone, aprepitant, bexarotene, clarithromycin, itraconazole, ketoconazole, St. John's wort).
10. Patients who have chronic active hepatitis.
11. Patients taking any of the following medications who cannot discontinue these medications for three months during administration of ketoconazole; statin cholesterol medications, cyclosporine, isoniazid, rifampin, terfenadine, triazolam or astemizole.
12. Patients who have history of cerebrovascular accident, deep venous thrombosis, pulmonary emboli, unstable angina or clinical congestive heart failure.
13. Medical conditions, which, in the opinion of the investigators would jeopardize either the patient or the integrity of the data obtained.
14. Patients unwilling to use contraceptives while on study.
15. Patients with a risk of nodal involvement of greater than 10% should have received a bone scan and CT of the pelvis prior to screening for the study as part of standard of care.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-07; Primary Completion 2010-06 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Bruce Montgomery, MD, Principal Investigator — University of Washington; Seattle Cancer Care Alliance; VA Puget Sound HCS; Peter S. Nelson, MD, Principal Investigator — Fred Hutchinson Cancer Research Center; Seattle Cancer Care Alliance
Locations (2):
- United States (2):
  - Veterans' Administration Puget Sound Health Care System (VAPSHCS), Seattle, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Mostaghel EA, Nelson PS, Lange P, Lin DW, Taplin ME, Balk S, Ellis W, Kantoff P, Marck B, Tamae D, Matsumoto AM, True LD, Vessella R, Penning T, Hunter Merrill R, Gulati R, Montgomery B. Targeted androgen pathway suppression in localized prostate cancer: a pilot study. J Clin Oncol. 2014 Jan 20;32(3):229-37. doi: 10.1200/JCO.2012.48.6431. Epub 2013 Dec 9. PMID 24323034
- [Derived] Tamae D, Byrns M, Marck B, Mostaghel EA, Nelson PS, Lange P, Lin D, Taplin ME, Balk S, Ellis W, True L, Vessella R, Montgomery B, Blair IA, Penning TM. Development, validation and application of a stable isotope dilution liquid chromatography electrospray ionization/selected reaction monitoring/mass spectrometry (SID-LC/ESI/SRM/MS) method for quantification of keto-androgens in human serum. J Steroid Biochem Mol Biol. 2013 Nov;138:281-9. doi: 10.1016/j.jsbmb.2013.06.014. Epub 2013 Jul 10. PMID 23851165
- [Derived] Dean JP, Sprenger CC, Wan J, Haugk K, Ellis WJ, Lin DW, Corman JM, Dalkin BL, Mostaghel E, Nelson PS, Cohen P, Montgomery B, Plymate SR. Response of the insulin-like growth factor (IGF) system to IGF-IR inhibition and androgen deprivation in a neoadjuvant prostate cancer trial: effects of obesity and androgen deprivation. J Clin Endocrinol Metab. 2013 May;98(5):E820-8. doi: 10.1210/jc.2012-3856. Epub 2013 Mar 26. PMID 23533230
- Available data/document: Paper with attached protocol and outcomes — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3887479/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 12 | 10 | 13
Completed | 12 | 10 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 12 | 10 | 13 | 35
Age, Continuous [Median (Full Range); unit: years] | 62 [41 to 82] | 66 [41 to 82] | 60 [41 to 82] | 64 [41 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 12 | 10 | 13 | 35
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 13 | 35

OUTCOME MEASURES:

1. Primary Outcome: Prostate Tissue DHT
Description: Tissue dihydrotesterone (DHT)
Time Frame: After 12 weeks of neoadjuvant androgen deprivation
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 12 | 10 | 13
ng/g | 0.03 (0.01) | 0.06 (0.06) | 0.03 (0.02)

2. Secondary Outcome: To Determine the Effects of Different Modes of Androgen Deprivation on Serum DHT
Description: Serum DHT
Time Frame: After 12 weeks of neoadjuvant androgen deprivation
Population: Patients with clinically localized prostate cancer treated for 3 months with the treatments in Groups 1-3
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 12 | 10 | 13
ng/dL | 4.2 (3.4) | 3.6 (2.0) | 5.7 (4.9)

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/13
Other Adverse Events (participants affected / at risk) | 12/12 | 10/10 | 13/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=12) | Group 2 (N=10) | Group 3 (N=13)
hot flushes (Vascular disorders) | 12 (12) | 10 (10) | 13 (13)
Fatigue (General disorders) | 5 (5) | 6 (6) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No